CLINICAL TRIAL: NCT01099852
Title: Descriptive and Prognostic Study of Arbovirus Infections in France, Based on a Hospital Cohort of Children and Adults With Suspected Arbovirose.
Brief Title: Cohort of Patients Infected by an Arbovirus
Acronym: CARBO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Clinique Antilles-Guyane (Other)
Responsible Party: Sponsor
Other Study IDs: 09/B/08
Record Dates: First submitted 2010-02-23; First posted 2010-04-08 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Fever; Dengue; Chikungunya; Zika Virus
Keywords: dengue; fever; dengue hemorrhagic fever; dengue virus; Chikungunya virus; Zika Virus; Joint pain
MeSH Terms: conditions — Fever; Dengue; Chikungunya Fever; Zika Virus Infection; Severe Dengue; Arthralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, plasma, DNA, Urine
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: biological sample collection — blood sample collection urine sample cerebrospinal fluid sample
Other: Quality of life Questionnaire EuroQol® — Changes in quality of life, measured with the EuroQol® questionnaire 3 and 12 weeks after the onset of dengue fever symptoms.
Other: Health Assessment Questionnaire - MDHAQ and RAPID3 — Questionnaire used at the 3rd month of follow up.
Other: Neuropathic Pain Questionnaire (DN4) — Questionnaire used during the follow up

SUMMARY:
There are hundred of arbovirus which have been shown to cause disease in humans. Their most common clinical symptoms are algo-eruptive (dengue, chikungunya, zika), hemorrhagic fever (dengue, yellow fever, Crimean-Congo hemorrhagic fever), neurological (West Nile, Zika, dengue, Japanese encephalitis) or arthritic afflictions (Chikungunya, O'nyong nyong). Dengue is a mosquito-born viral disease caused by 4 different serotypes of virus. Dengue fever (DF) is defined by the sudden onset of fever with non-specific constitutional symptoms, recovery occurring spontaneously in 3 to 7 days. The infection can sometimes progress to dengue hemorrhagic fever (DHF) characterized by a transient increase in vascular permeability provoking a plasma leakage syndrome. DHF can be complicated by shock and internal hemorrhage. Other rarer complications include encephalitis, hepatitis, rhabdomyolysis and myocarditis. There is currently no way of predicting the outcome of DF or DHF and the WHO classification lacks sufficient sensitivity and specificity to recognize and guide the management of severe forms of dengue. The pathophysiology of these forms is also poorly known. Since 2000s, the French West Indies and Guiana have become hyperendemic for dengue with simultaneous circulation of the 4 serotypes, regular large outbreaks and severe dengue including fatalities. Chikungunya is a re-emerging virus causing massive epidemics in Africa, in the Indian Ocean and Southeast Asia. The first autochthonous cases were described in French Antilles in Nov 2013. The disease typically consists of an acute illness like dengue fever with abrupt onset of a high-grade fever followed by constitutionals symptoms, poly-arthritis and skin involvement. Usually, the illness resolves in 4 to 6 weeks. However, severe clinical forms in early stage may appear and chronic clinical forms as incapacitating arthralgia which affect 40 to 60% of patients. In France, others arboviruses may cause severe emerging and re-emerging infectious diseases like Zika or West Nile. In non-immunized population these emerging diseases may cause outbreaks with specific severe clinical complications. The French interministerial mission on emerging infectious diseases coordinated by Professor Antoine Flahault, recommended such studies: large prospective multicenter cohort studies to characterize severe forms of arbovirus infections to seek predictive factors and to investigate the pathophysiology of the diseases.

DETAILED DESCRIPTION:
Principal objective To identify demographic, clinical, biological, virologic, immunologic and genetic factors associated with or predictive of severe complications of arbovirus infections (shock, internal bleeding, organ failure, death) in a cohort of children and adults with confirmed arbovirus infections, in France.

Secondary objective

To identify demographic, clinical, biological, virologic, immunologic and genetic factors predictive of altered quality of life after confirmed an acute arbovirus infection. Onset of specific complications:

* Hemorrhagic fever (dengue: WHO criteria)
* Neurological disorders (West Nile virus infection, Zika virus infection, Japanese encephalitis…)
* Chronic chikungunya (persistent Chronic chikungunya (persistent musculoskeletal symptoms for more than three months after symptoms onset)

ELIGIBILITY:
INCLUSION CRITERIA :

* Adult, child or newborn with a weight > 2.5 kg the days of enrollment.
* Consulting a participating hospital center (emergency room, full hospitalization, day hospitalization, or outpatient visit).
* Arbovirosis suspected or confirmed biologically: A suspected case of arbovirus infection is defined by:

  * The combination of clinical and biological signs observed suggestive of arbovirosus infection: fever (reported by the patient or family, or documented), headache, rash, myalgia, arthralgia, abdominal pain, hemorrhage, thrombocytopenia, or
  * Children under 6 years: the report (by family or documented) of a fever on the day of enrollment or within 7 previous days, possibly accompanied by a of pain - At a patient with a notion of stay in 2 weeks preceding in a zone of arbovirus circulation (only for the imported cases)

A case of arbovirus infection confirmed biologically is defined by:

* RT-PCR arbovirus positive in plasma or urine (Zika virus infection), or by detection of the NS1 antigen (dengue), or an appearance or an significant increase (multiplication of the title by four) of the G immunoglobulin directed against arbovirus in question on an early taken serum (during the first week following the start of symptoms) and another taken at least 10 days later.
* Symptom onset within the 7 days before the enrollment visit or within 21 days for severe forms of the disease.Possibility of follow-up throughout study period. * Acceptance to participate in the study and in follow-up; informed consent of the patient (adult and minor in age to express his desire) or a legal representative (for minors, and patients unable to sign the consent form).

EXCLUSION CRITERIA :

* No follow-up possible after the first visit
* Patient or holder of parental authority not registered in the French medical social security national program

Min Age: 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital cohort of children and adults with suspected of infectious by an arbovirus in the overseas departments and regions and in France.
Sampling Method: Non-Probability Sample
Enrollment: 1377 (Estimated)
Dates: Start 2010-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence, during follow-up (for 12 weeks following symptom onset), of shock, internal bleeding, failure of one or several organs or systems (brain, heart, lung, liver, kidney, clotting system), or death. | 12 weeks
  The primary endpoint is a composite endpoint defined as the occurrence, within 12 weeks of the onset of arbovirosis, of at least 1 of the following events: death or shock or internal bleeding, or failure to one or more organs or systems (brain, heart, lung, liver, kidney, hemostasis). Deaths not attributable directly or indirectly to the arbovirosis in question will not be taken into account.

SECONDARY OUTCOMES:
Specific complications: Onset of hemorrhagic fever (dengue) Onset of encephalitis or neurological disorders (West Nile virus, Japanese encephalitis, Zika virus) Onset of chronic form (Chikungunya) | 12 weeks
  The analysis will focus only on patients with biologically confirmed arbovirosis by one of the following exams:
  * RT-PCR plasma (arbovirus), or urine (Zika virus),
  * Research of the NS1 positive antigen (dengue),
  * Significant appearance or increase of the G immunoglobulin directed against the arbovirus in question between an early serum (during the first week following the onset of symptoms) and another taken at least 10 days later

CONTACTS AND LOCATIONS:
Overall Officials: Andre Cabie, MD, Principal Investigator — CHU de Martinique
Locations (8):
- France (3):
  - Hôpital Saint André, Bordeaux
  - Hôpital La Pitié Salpêtrière, Paris
  - Hôpital Bichat-Claude Bernard, Paris
- CH André Rosemond, Cayenne, French Guiana
- CHU de Pointe à Pitre/Abymes, Pointe-à-Pitre, Guadeloupe
- Centre Hospitalier Universitaire de Martinique, Fort-de-France, Martinique
- Reunion (2):
  - CHU de la Réunion, Saint-Denis
  - Centre Hospitalier Gabriel Martin, Saint-Paul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carras M, Maillard O, Cousty J, Gerardin P, Boukerrou M, Raffray L, Mavingui P, Poubeau P, Cabie A, Bertolotti A. Associated risk factors of severe dengue in Reunion Island: A prospective cohort study. PLoS Negl Trop Dis. 2023 Apr 17;17(4):e0011260. doi: 10.1371/journal.pntd.0011260. eCollection 2023 Apr. PMID 37068115
- [Derived] Bertolotti A, Thioune M, Abel S, Belrose G, Calmont I, Cesaire R, Cervantes M, Fagour L, Javelle E, Lebris C, Najioullah F, Pierre-Francois S, Roze B, Vigan M, Laouenan C, Cabie A; Chronic Chikungunya working group of University Medical Center of Martinique. Prevalence of chronic chikungunya and associated risks factors in the French West Indies (La Martinique): A prospective cohort study. PLoS Negl Trop Dis. 2020 Mar 12;14(3):e0007327. doi: 10.1371/journal.pntd.0007327. eCollection 2020 Mar. PMID 32163420